CLINICAL TRIAL: NCT04257630
Title: Influence of Coping Strategies on Short and Long-term Outcomes of Pulmonary Rehabilitation in Patients With Idiopathic Pulmonary Fibrosis (IPF) and Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Coping Strategies Within Pulmonary Rehabilitation in Patients With IPF and COPD
Status: Completed | Type: Observational
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Professor for pulmonary rehabilitation, Schön Klinik Berchtesgadener Land
Other Study IDs: PsyLu-Study
Record Dates: First submitted 2020-01-28; First posted 2020-02-06 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Idiopathic Pulmonary Fibrosis; Chronic Obstructive Pulmonary Disease
Keywords: coping strategies; psychological burden; anxiety; depression; quality of life; pulmonary rehabilitation
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Disease, Chronic Obstructive; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this prospective observational trial is to evaluate the influence of Coping strategies on pulmonary rehabilitation outcomes like 6-minute walk distance and Quality of life.

DETAILED DESCRIPTION:
In the recent pulmonary rehabilitation (PR) statement of the American Thoracic Society/ European Respiratory Society, PR is mentioned to be beneficial by improving exercise capacity, symptoms and quality of life in patients with other chronic respiratory diseases than chronic obstructive pulmonary disease (COPD) (1). Although patients with idiopathic pulmonary fibrosis (IPF) often suffer from psychological distress such as symptoms of anxiety and depression, only little is known about the impact of these mental co-morbidities on PR outcomes.

In a former study the investigators demonstrated that patients with IPF benefit well from an inpatient PR program of only 3 weeks duration by improving exercise capacity (6-Minute walk distance), health-related quality of life as well as symptoms of anxiety and depression. During the 3-months follow-up after PR, most of these improvements disappeared so that this group showed similar values at follow-up compared to baseline. However, in contrast patients from the control-group with usual care worsened significantly during the 6 months study period.

Interestingly, a linear regression analysis revealed that IPF patients with lower levels of anxiety showed the tendency to have the best sustainability in exercise capacity at the 3 months follow-up. Given that maintenance of exercise capacity may be crucial to influence prognosis and the risk of mortality, reducing symptoms of anxiety might be of special interest.

The negative influence of anxiety symptoms on exercise capacity is a new finding in IPF patients but already known in the field of other chronic diseases: in patients with chronic pain and recently also in patients with COPD, "fear avoidance" behavior is discussed as having a direct negative influence on daily physical activity levels. COPD patients seem to develop fear/anxiety of exercise-related dyspnea due to classical and operant conditioning. This may lead to consecutive avoidance of physical activity and other exercises in daily life (2).

Anxiety symptoms and psychological distress have been shown to be related to patients individual illness perceptions and their way of coping with the disease like e.g. problem-focusing coping, looking for information, depressive coping.

In patients with IPF, the role of coping styles in the context of PR has not been investigated yet. It is unclear whether anxiety symptoms are influenced by individual characteristics of IPF patients such as specific coping strategies and illness perceptions and therefore, whether individual coping strategies might have an influence on the PR outcome.

This latter might be an underestimated issue influencing the PR effects in patients with chronic respiratory diseases. Better knowledge in this field is of special clinical importance in order to ensure short- und long term PR success. Potential differences in psychological profiles or coping strategies between COPD and IPF patients might result in disease-specific interventions during and after PR.

Therforme, aim of this study is to evaluate the influence of coping strategies on pulmonary rehabilitation outcomes.

This study is a prospective observational trial. Asssessments will take place at admission of the rehabilitation program, at discharge and partially after 3-month.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic pulmonary fibrosis with a FVC between 30 to 70% predicted or
* Patients with chronic obstructive pulmonary disease (GOLD stage III and IV)
* Age: 50-80 years
* Medical treatment according to recent guidelines (including long-term oxygen therapy and or non invasive ventilation)
* Written informed consent

Exclusion Criteria:

* General exclusion criteria for physical training like acute coronary syndrome, acute myo- or pericarditis, acute lung embolism, acute heart failure or orthopedic co-morbidities which prevent patients from participating in training program
* Non-compliance

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who take part in a pulmonary rehabilitation program at Schoen Klinik Berchtesgadener land will recruited.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Coping strategies in anxious vs. non-anxious IPF-patients | Day 1, Day 21 and 3-months after pulmonary rehabilitation program (Day 21)
  Difference in Essener Coping questionnaire in axious (Hospital anxiety and Depression scale [HADS]>=8points) and non-anxious (HADS<8points) IPF-patients

SECONDARY OUTCOMES:
Correlation between 6-minute walk distance and Essener Coping questionnaire | Day 1 and Day 21
  The essener Coping questionnaire measures coping mechanisms; a 45-item self-report questionnaire; higher scores indicate higher presence of the respective state
Correlation between Health related Quality of life and Essener Coping questionnaire | Day 1, Day 21 and 3-months after pulmonary rehabilitation program
  Health related Quality of life will be assessed by chronic respiratory disease questionnaire (CRQ)- a 20-item self-report questionnaire; score 1-7; higher scores indicate a better health-related quality of life
  ; The essener Coping questionnaire measures coping mechanisms; a 45-item self-report questionnaire; higher scores indicate higher presence of the respective state
Correlation between 6-minute walk distance and Hospital Anxiety and Depresion scale | Day 1 and Day 21
  Anxiety/Depression measured by Hospital Anxiety and Depression Scale (HADS) - a screening questionnaire including 6 questions about depression and 8 questions about anxiety; higher scores indicate higher presence of anxiety/ depression
Correlation between 6-minute walk distance and COPD anxiety questionnaire | Day 1 and Day 21
  assessed by the German "COPD Angst Fragebogen" (CAF) - a 20-item self-report questionnaire, rated on a Lickert-scale (score 0-4); maximum score: 80 points; higher scores indicate higher anxiety levels.
Correlation between 6-minute walk distance and Illness Perception Questionnaire | Day 1 and Day 21
  assessed by the Illness perception Questionnaire, revised (IPQ-R) - 18 items, score 1-5; higher scores indicate a worse illness perception, except of item 7,9,10,11,12.
Correlation between 6-minute walk distance and Patient-Health questionnaire | Day 1 and Day 21
  Depression measured by Patient-Health questionnaire including 9 items; each question range from 0 to 3; higher scores indicate higher presence of the respective state
Correlation between 6-minute walk distance and Health related Quality of life | Day 1 and Day 21
  Health related Quality of life will be assessed by chronic respiratory disease questionnaire (CRQ)- a 20-item self-report questionnaire; score 1-7; higher scores indicate a better health-related quality of life
Correlation between 6-minute walk distance and SF-36 survey | Day 1 and Day 21
  Health related quality of life will be measured by SF-36 questionnaire; a screening questionnaire including 36-items; higher score indicate higher quality of life
Correlation between 6-minute walk distance and King´s Brief Interstitial lung disease questionnaire | Day 1 and Day 21
  Health Status measured by King's Brief Interstitial lung disease questionnaire including 15 items; higher scores indicate better respective state
Correlation between physical activity level and Essener Coping questionnaire | 2 weeks and 3 months after pulmonary rehabilitation program completion (Day 21) activity monitoring for 5 week days each
  The essener Coping questionnaire measures coping mechanisms; a 45-item self-report questionnaire; higher scores indicate higher presence of the respective state
Correlation between physical activity level and Hospital Anxiety and Depresion scale | 2 weeks and 3 months after pulmonary rehabilitation program completion (Day 21) activity monitoring for 5 week days each
  Anxiety/Depression measured by Hospital Anxiety and Depression Scale (HADS) - a screening questionnaire including 6 questions about depression and 8 questions about anxiety; higher scores indicate higher presence of anxiety/ depression
Correlation between physical activity level and COPD anxiety questionnaire | 2 weeks and 3 months after pulmonary rehabilitation program completion (Day 21) activity monitoring for 5 week days each
  assessed by the German "COPD Angst Fragebogen" (CAF) - a 20-item self-report questionnaire, rated on a Lickert-scale (score 0-4); maximum score: 80 points; higher scores indicate higher anxiety levels.
Correlation between physical activity level and Illness Perception Questionnaire | 2 weeks and 3 months after pulmonary rehabilitation program completion (Day 21) activity monitoring for 5 week days each
  assessed by the Illness perception Questionnaire, revised (IPQ-R) - 18 items, score 1-5; higher scores indicate a worse illness perception, except of item 7,9,10,11,12.
Correlation between physical activity level and Patient-Health questionnaire | 2 weeks and 3 months after pulmonary rehabilitation program completion (Day 21) activity monitoring for 5 week days each
  Depression measured by Patient-Health questionnaire including 9 items; each question range from 0 to 3; higher scores indicate higher presence of the respective state
Correlation between physical activity level and chronic respiratory disease questionnaire | 2 weeks and 3 months after pulmonary rehabilitation program completion (Day 21) activity monitoring for 5 week days each
  Depression measured by Patient-Health questionnaire including 9 Items; each question range from 0 to 3; higher scores indicate higher presence of the respective state
Correlation between physical activity level and SF-36 survey | 2 weeks and 3 months after pulmonary rehabilitation program completion (Day 21) activity monitoring for 5 week days each
  Health related quality of life will be measured by SF-36 questionnaire; a screening questionnaire including 36-items; higher score indicate higher quality of life
Correlation between physical activity Level and King´s Brief Interstitial lung disease questionnaire | 2 weeks and 3 months after pulmonary rehabilitation program completion (Day 21) activity monitoring for 5 week days each
  Health Status measured by King's Brief Interstitial lung disease questionnaire including 15 items; higher scores indicate better respective state
Differences in Coping mechanisms between IPF and COPD patients | Day 1, Day 21 and 3-months after pulmonary rehabilitation program (Day 21)
  The essener Coping questionnaire measures coping mechanisms; a 45-item self-report questionnaire; higher scores indicate higher presence of the respective state

CONTACTS AND LOCATIONS:
Locations (1):
- Schoen Klinik BGL, Schoenau Am Königssee, Bavaria, Germany

REFERENCES:
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Hallas CN, Howard C, Theadom A, Wray J. Negative beliefs about breathlessness increases panic for patients with chronic respiratory disease. Psychol Health Med. 2012;17(4):467-77. doi: 10.1080/13548506.2011.626434. Epub 2012 Feb 13. PMID 22329594